CLINICAL TRIAL: NCT03656016
Title: Assessment of Cerebrospinal Fluid Flow Related Disorders Using a Phase-contrast Magnetic Resonance Imaging Technique.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shimaa Hassanien Hassanien Bakr, principal Investigator, Assiut University
Other Study IDs: CSFFPCMRI
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-01

CONDITIONS: Cerebrospinal Fluid
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- study group: patients with congenital and acquired disorders that can alter the CSF dynamics will undergo phase-contrast magnetic resonance imaging
  Interventions: Device: Magnetic Resonance Imaging
- control group: age matched healthy individuals will undergo phase-contrast magnetic resonance imaging
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Phase contrast magnetic resonance imaging technique

SUMMARY:
Cerebrospinal fluid is a clear, colorless fluid that circulates in the cranial and spinal subarachnoid spaces, located between the pia and arachnoid matters. It is mainly produced by the choroid plexus, while lesser amount produced by the ependymal cells lining the ventricles. Its function includes cushioning and lubrication of the central nervous system, circulation of nutrients and waste collection providing basic mechanical and immunological protection to the brain.

DETAILED DESCRIPTION:
There are several disorders such as communicating and non- communicating hydrocephalus, normal pressure hydrocephalus, cystic cerebrospinal fluid collections, Chiari malformation, syringomyelic cyst and arachnoid cyst that can change the cerebrospinal fluid dynamics.

Rapid advances in imaging techniques have remarkably improved the diagnosis and treatment of these disorders.

Phase contrast magnetic resonance imaging is a rapid, simple and non-invasive technique which is sensitive to even small cerebrospinal fluid flows, and can be used to evaluate cerebrospinal fluid flow both qualitatively and quantitatively. Cine phase contrast magnetic resonance images show cerebrospinal fluid flow in a dynamic, more easily appreciable, and in a more pleasing manner, allowing the delineation of obstruction, if present, along the portions of cerebrospinal fluid pathway where obstruction is common.

Phase contrast magnetic resonance imaging can be used to discriminate between communicating hydrocephalus and non-communicating hydrocephalus, to localize the level of obstruction in obstructive hydrocephalus, to determine whether arachnoid cysts communicate with the subarachnoid space, to differentiate between arachnoid cysts and subarachnoid space, to discriminate between syringomyelia and cystic myelomalacia, and to evaluate flow patterns of posterior fossa cystic malformations.

This imaging method can also provide significant information in pre-operative evaluation of Chiari 1 malformation and post-operative follow-up of patients with neuroendoscopic third ventriculostomy and ventriculoperitoneal shunt.

The application of cine phase contrast magnetic resonance imaging technique in patients with normal pressure hydrocephalus holds great promise for improvement of the diagnosis, especially in those cases where the differentiation from atrophy on clinical and conventional radiological basis is difficult.

ELIGIBILITY:
Inclusion Criteria:

* Patients with different age groups and both sex with clinical and routine conventional magnetic resonance imaging findings suggestive of cerebrospinal fluid flow disorders.

Exclusion Criteria:

1. Patients with contraindications for MRI, e.g. an implanted magnetic device, pacemakers or claustrophobia.
2. Patients with VP shunts
3. Patients with ventriculomegally due to brain SOLs.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with different age groups and both sex with clinical and routine conventional magnetic resonance imaging findings suggestive of cerebrospinal fluid flow disorders
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To calculate different cerebrospinal fluid flow parameters at different levels of flow quantification. | base line
  measure Systolic stroke volume and Peak systolic velocity at different levels of flow quantification

SECONDARY OUTCOMES:
To correlate these parameters to the normal values of age matched control group | baseline
  correlate Systolic stroke volume and Peak systolic velocity with normal values

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa Bakr, MSc, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sakka L, Coll G, Chazal J. Anatomy and physiology of cerebrospinal fluid. Eur Ann Otorhinolaryngol Head Neck Dis. 2011 Dec;128(6):309-16. doi: 10.1016/j.anorl.2011.03.002. Epub 2011 Nov 18. PMID 22100360
- [Background] Yildiz H, Yazici Z, Hakyemez B, Erdogan C, Parlak M. Evaluation of CSF flow patterns of posterior fossa cystic malformations using CSF flow MR imaging. Neuroradiology. 2006 Sep;48(9):595-605. doi: 10.1007/s00234-006-0098-8. Epub 2006 Jun 3. PMID 16752134
- [Background] Yamada S, Tsuchiya K, Bradley WG, Law M, Winkler ML, Borzage MT, Miyazaki M, Kelly EJ, McComb JG. Current and emerging MR imaging techniques for the diagnosis and management of CSF flow disorders: a review of phase-contrast and time-spatial labeling inversion pulse. AJNR Am J Neuroradiol. 2015 Apr;36(4):623-30. doi: 10.3174/ajnr.A4030. Epub 2014 Jul 10. PMID 25012672
- [Background] Parkkola RK, Komu ME, Aarimaa TM, Alanen MS, Thomsen C. Cerebrospinal fluid flow in children with normal and dilated ventricles studied by MR imaging. Acta Radiol. 2001 Jan;42(1):33-8. doi: 10.1080/028418501127346431. PMID 11167329
- [Background] Ng SE, Low AM, Tang KK, Lim WE, Kwok RK. Idiopathic normal pressure hydrocephalus: correlating magnetic resonance imaging biomarkers with clinical response. Ann Acad Med Singap. 2009 Sep;38(9):803-8. PMID 19816640